CLINICAL TRIAL: NCT04527276
Title: Reducing the Incidence of Ventilator Associated Pneumonia in Critically Ill Children: a Randomized Controlled Trial to Assess the Efficacy of Oral Mucosal Mouthwashes With Chlorhexidine
Brief Title: Reducing the Incidence of VAP in Critically Ill Children and Assessment of Oral Care With CHX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Zeynep Karakaya, Principal investigator, Istanbul Medeniyet University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IstanbulIMU
Record Dates: First submitted 2020-08-17; First posted 2020-08-26 (Actual); Last update posted 2020-08-26 (Actual); Status verified 2020-08

CONDITIONS: Ventilator Associated Pneumonia
Keywords: Oral care; Chlorhexidine; ventilator associated pneumonia
MeSH Terms: conditions — Pneumonia, Ventilator-Associated

STUDY DESIGN:
Intervention Model Description: All patients were consecutively randomized (1:1) to receive either 0.12% CHX rinse solution or placebo applications using a computer generated balanced randomization table.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chlorhexidine (Active Comparator): 5 ml of 0,12 % Chlorhexidine (CHX) solution is applied to the intervention group for oral care
  Interventions: Other: Oral care with 0,12% Chlorhexidine
- Placebo Group (No Intervention): Group of patients who received standard oral care

INTERVENTIONS:
Other: Oral care with 0,12% Chlorhexidine — 0, 12 % CHX, and standard oral care with 0,9% NaCl were compared to assess VAP rates. Both solutions were applied to critically ill children who were intubated.
  Arms: Chlorhexidine

SUMMARY:
This was a single-centered, randomized, placebo-controlled double-blind clinical trial conducted in the pediatric intensive care unit (PICU), in patients who were aged 1 month to 18 years, needing MV for at least 48 hours, to evaluate the effect of Chlorhexidine (CHX) on Ventilator-associated pneumonia (VAP) incidence and to determine VAP risk factors.

DETAILED DESCRIPTION:
Patients were randomized into two groups receiving CHX (0.12%) or placebo (0.9% NaCl) and followed for VAP development. All patients were consecutively randomized (1:1) to receive either 0.12% CHX rinse solution or placebo applications using a computer generated balanced randomization table. The unlabeled standardized tubes containing placebo or 0.12% CHX were serially numbered and bagged for each patient according to randomization. The preparation of bagged treatments and their numbering were done by the same personnel who was not involved in the study. The placebo rinse contained 0.9% NaCl (normal saline [NS]), and was identical to the 0.12% CHX rinse solution with regard to appearance, consistency, taste and smell. The patients, physicians, outcome assessors, and data analysts were kept blinded to the intervention.

The standard care protocols in the PICU were performed. Before beginning the study, nurses received a training program for VAP prevention, procedure/technique for oral hygiene and use of oral mucosa assessment score under supervision of pediatric residents. They were trained on the method of application of solutions according to CDC guidelines in order to ensure uniform treatments. Nurses were double blinded and had no knowledge of the solution they were using.

Both treatment groups (placebo and 0.12% CHX) received treatments at 4-hour intervals, nurses used the whole content of 5 ml tubes containing rinse solution. In both groups, nurses performed oral cleansing as follows: first, the endotracheal cuff pressure was tested to ensure proper pressure prior to oral care and oropharyngeal secretions were aspirated to remove any accumulated secretions. Then the application of rinse solutions to cleanse all areas of the oral cavity, including the anterior and posterior pharynx, gums, teeth, tongue, and buccal mucosa, with standard disposable applicator (foam swab) was applied, followed by removal of excess solution from the mouth by a sterile catheter. Strict hand hygiene was ensured during the procedures. The period of application was from the day of intubation until extubation. Presence of any adverse effect of the solutions was recorded. Beck oral assessment score (BOAS) was used twice daily to evaluate the oral health of both groups.

ELIGIBILITY:
Inclusion Criteria:

* aged 1 month to 18 years
* needing MV for at least 48 hours
* PICU patients

Exclusion Criteria:

* not consenting to participate in the study
* known hypersensitivity to CHX
* presence of tracheotomy,
* undergoing MV for less than 48 hours
* having received MV for more than 24 hours prior to PICU admission
* readmission to PICU
* suspected or diagnosed immunodeficiency
* history of malignant disease(active or at remission),
* being diagnosed with oral mucositis or periodontal disease
* chronic pulmonary and/or cardiac diseases
* having severe oral/facial trauma,
* use of immunosuppressive drugs (such as corticosteroids).

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 138 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Prevalance of VAP | 14 days
  Prevalance of VAP /1000 ventilator days (actual number of VAP episodes)
Characteristics of VAP | 14 days
  Early onset vs. late onset VAP rate

SECONDARY OUTCOMES:
Causative organisms of VAP | 14 days
  Type of micro-organisms causing VAP in both groups
Duration of PICU stay | 12 months
  Median duration of PICU stay (days)
Duration of Hospital stay | 12 months
  Median duration of hospital stay (days)
Duration of ventilation | 12 months
  Median duration of mechanical ventilation (days)
Survival | 12 months
  Rate of survival
Causative organism of VAP | 14 days
  number of microorganism
Causative organism | 14 days
  percentage of microorganism causing VAP

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medeniyet University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Karakaya Z, Duyu M, Yersel MN. Oral mucosal mouthwash with chlorhexidine does not reduce the incidence of ventilator-associated pneumonia in critically ill children: A randomised controlled trial. Aust Crit Care. 2022 Jul;35(4):336-344. doi: 10.1016/j.aucc.2021.06.011. Epub 2021 Aug 8. PMID 34376358